CLINICAL TRIAL: NCT01663077
Title: Clozapine Fixed Dose Steady State Plasma Levels and the Relationship to the Polymorphism of CYP1A2, CYP3A4, CYP3A5 and CYP2D6 in Clinically Stable Schizophrenic Adult Patients
Brief Title: Clozapine Plasma Levels and the Relationship to the Genetic Polymorphism in Shizophrenic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tirat Carmel Mental Health Center (Other Government)
Collaborators: Technion, Israel Institute of Technology (Other); Ben-Gurion University of the Negev (Other); Beersheva Mental Health Center (Other Government); Sha'ar Menashe Mental Health Center (Other); HaEmek Medical Center, Israel (Other); The Nazareth Hospital, Israel (Other)
Responsible Party: Principal Investigator, Anatoly Kreinin, MD, PHD, Director of Psychiatric Department, Tirat Carmel Mental Health Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KBK2012; 03/11 (Other: Tirat Carmel Mental Health Center Review Board)
Record Dates: First submitted 2012-07-25; First posted 2012-08-13 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Schizophrenia
Keywords: Clozapine; Schizophrenia; Remissia; polymorphism
MeSH Terms: conditions — Schizophrenia | interventions — Clozapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clozapine (Experimental): Clozapine tablet 150 mg at the day and 150 mg in the evening by mouth per day for 3 month
  Interventions: Drug: Clozapine

INTERVENTIONS:
Drug: Clozapine — A fixed dose of Clozapine 300 mg/day (150 mg x 2)for 3 month
  Other Names: Leponex

SUMMARY:
Approximately 30-60% of all schizophrenia patients who fail to respond to typical antipsychotics may respond to Clozapine. Clozapine has long been considered the "gold standard" within the atypical neuroleptic spectrum, backed by years of clinical experience and research, but uncertainties remain in some aspects of this drug. One such question is the link between dose, blood levels and patient clinical response. The Clozapine therapeutic plasma levels range between 250 - 450 ng/mL creating difficulties in using these results in routine clinical practice. Approximately 30% - 51% of "treatment-resistant schizophrenia" patients do not fully respond to Clozapine, a poorly understood phenomenon. Factors relevant to Clozapine-resistance include co-morbidity, drug misuse, poor adherence, inadequate duration of treatment and inadequate dose/plasma-levels. Pharmacogenetic factors such as different polymorphisms in involved genes may play a role. Pharmacodynamic and genetic data appear important in determining the clinical response to Clozapine. Clozapine-treated patients possessing different 3A4 polymorphisms, may respond differently as compared to other patients having normal 3A4 alleles. Recently, the CYP2D6 has also been involved in this drug metabolic pathway. Population pharmacokinetics of clozapine evaluated with the nonparametric maximum likelihood method. This pharmacogenetic explanation/hypothesis may explain Clozapine- resistance in schizophrenics.

The high variability in plasma levels requires a large study in order to be able to determine correlation between clinical efficacy and plasma levels and genotyping. A preliminary study will enable power analysis and adequate determination of sample size.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV criteria for schizophrenia (American Psychiatric Association 2000)
* All clozapine mono-therapy patients (only 300 mg/day) who respond to treatment and achieved symptomatic remission (45, 46) and were stable for at least 3 month will be included
* No change in benzodiazepine medications for the trial period.
* Legal ability and willingness to sign an informed consent form for participation in the study.

Exclusion Criteria:

* Evidence of serious neurologic or endocrine disorder, for example severe head trauma, seizure disorder, dementia, Cushing's disease, thyroid disorder, mental retardation, alcohol or drug abuse, substance dependence (other than nicotine dependence), or presenting symptoms likely substance- induced, as judged by a study physician.
* Unstable medical illness or neurologic illness (seizures, CVA); breast, uterine, or ovarian cancer.
* Pregnant women, use of oral contraceptives or other hormonal supplementation such as estrogen. [Female patients will also have a pregnancy test.].

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Clozapine steady state plasma level | 3 month

SECONDARY OUTCOMES:
Polymorphism of CYP1A2, CYP3A4, CYP3A5 and CYP2D6 in clinically stable schizophrenic adult patients | Once

CONTACTS AND LOCATIONS:
Overall Officials: Anatoly Kreinin, MD, Phd, Study Director — Tirat Carmel Mental Health Center; Yedidia Bentur, MD, Principal Investigator — Rambam Health Care Campus, Haifa; Norberto Krivoy, MD, Principal Investigator — Rambam Health Care Campus, Haifa; David Rabinowitz, MD, Principal Investigator — Rambam Health Care Campus, Haifa; Kamal Farhat, MD, Principal Investigator — The Nazareth Hospital-EMM; Vladimir Lerner, MD, Phd, Principal Investigator — Beersheva Mental Health Center; Boaz Bloch, MD, Principal Investigator — Haemek Hospital, Afula; Alexander Grinshpoon, MD, MHA, PhD, Principal Investigator — Shaar Menashe MHC
Locations (1):
- Tirat Carmel Mental Health Center, Tirat Carmel, Israel